CLINICAL TRIAL: NCT06897514
Title: External Validation of Prediction Algorithm Using Non-invasive Monitoring Device for Intraoperative Hypotension
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Medical Center, Sungkyunkwan University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Professor, Anesthesiologist, Samsung Medical Center
Other Study IDs: SMC 2025-02-006
Record Dates: First submitted 2025-03-25; First posted 2025-03-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypotension During Surgery
Keywords: intraoperative hypotension; prediction algorithm
MeSH Terms: interventions — Prediction Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group (single group): All participants are enrolled in single group.
  Interventions: Diagnostic Test: Prediction algorithm for intraoperative hypotension

INTERVENTIONS:
Diagnostic Test: Prediction algorithm for intraoperative hypotension — All participants will receive five non-invasive monitoring during their surgery. Data from these monitoring device will be put into the prediction algorithm.

SUMMARY:
The goal of this prospective observational study is to externally validate the prediction algorithm using non-invasive monitoring device for intraoperative hypotension. The main question it aims to answer is: Does the prediction algorithm predict intraoperative hypotension effectively?

DETAILED DESCRIPTION:
The hypotension that occurs during surgery is associated with the poor prognosis of patients after surgery. Previous studies have reported that even a short period of time of hypotension increases the risk of postoperative complications such as kidney injury. If anesthesiologists can predict intraoperative hypotension in advance, they can prevent or minimize the damage.

Recently, there are many reports on medical artificial intelligence models that predict the intraoperative hypotension. Among them, the Hypotension Prediction Index (HPI) model has already been commercialized and used in clinical practice. However, HPI has limitations in that it is necessary to perform invasive techniques (arterial cannulation) or to use dedicated equipment at high cost. However, since many of the general anesthesia are performed without invasive monitoring devices, the use of HPI medical devices is subject to considerable restrictions.

The investigators have reported the prediction algorithm for intraoperative hypotension using five non-invasive monitoring devices commonly used in general anesthesia: 1) blood pressure (NBP, number), 2) electrocardiogram (ECG, waveform), 3) end-oxygen saturation waveform (PPG, waveform), 4) end-stage carbon dioxide waveform (ETCO2, waveform), and 5) an anesthesia depth (BIS, number) By conducting a retrospective external validation process using public clinical data from other institutions (tertiary hospital in Korea), the final model was able to have good predictability with an Area Under the Receiver-Operating Characteristic Curve (AUROC) value of 0.917.

However, investigators did not externally validate that algorithm through a prospective designed study. This study intends to externally validate the "hypertension prediction model during surgery using non-invasive monitoring device", which has already reported It is expected that the usefulness and limitations of the prediction model can be evaluated again, and the model can be advanced based on the results.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged 19 or more
* Elective surgery under general anesthesia
* American Society of Anesthesiologists physical status I - III

Exclusion Criteria:

* Vasopressor/Inotrope usage before surgery
* Patients who needs invasive arterial cannulation
* Emergency surgery
* Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who undergoing general anesthesia with five non-invasive monitoring device (non-invasive blood pressure, electrocardiography, photoplethysmography, capnography, and Bispectral Index)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Value of the Area Under the Receiver-Operating Characteristic curve analysis | 5 minutes before the occurrence of hypotension during general anesthesia
  The area under the receiver operating characteristic curve is a measurement of how well a prediction model can predict intraoperative hypotension. It is used to assess the performance of algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, MD PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong H, Kim D, Kim DW, Baek S, Lee HC, Kim Y, Ahn HJ. Prediction of intraoperative hypotension using deep learning models based on non-invasive monitoring devices. J Clin Monit Comput. 2024 Dec;38(6):1357-1365. doi: 10.1007/s10877-024-01206-6. Epub 2024 Aug 19. PMID 39158783